CLINICAL TRIAL: NCT04672148
Title: Prognostic Factors in Disease Progression and Mortality Risk in the Older Stroke Patients With Mechanical Thrombectomy
Brief Title: Prognostic Factors and Mortality in Older Stroke Patients With Mechanical Thrombectomy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 109125-E
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2020-12

CONDITIONS: Stroke, Ischemic
Keywords: Thrombectomy,acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Patient who died in the 30 days after receiving mechanical thrombectomy, no matter the mortality cause
- B: Non-30-day-mortality group after receiving mechanical thrombectomy

SUMMARY:
The study focus on the elderly patient (older than 80 years of age) who had acute ischemic stroke and received mechanical thrombectomy. The investigators analyze different factors in the stage of before, between, after procedure and trying to figure out if there is any difference between the 30-day-mortality group versus non-30-day-mortality group.

DETAILED DESCRIPTION:
With the constant improvements in health care, standard of living and the decrease birth rate, the percentage of the elderly population ( above 80 years old) is expected to double in Taiwan by the year 2044, according to data from the National Development Council. Consequently with the increase in the proportion of senior citizens, there will be an surge number of patient suffering from cardiovascular and cerebrovascular diseases, most importantly acute ischemic stroke. In recent years, mechanical thrombectomy has become the gold standard in the treatment for acute stroke patients, however, many studies have excluded the patients above the age of 80 years old as the benefits of the procedure have been very controversial and there is no clear evidence proving favorable a outcome. There are a few studies which state that though elderly patients had higher risk of complications when receiving mechanical thrombectomy as compared to younger patients, the prognosis was still superior to those didn't receive any intervention. Previous studies put more emphasis on the overall prognosis, morbidity and mortality rate, they didn't focused on the cause of mortality.

The study focuses on analyzing of the cause of mortality and whether there is a significant difference between 30-day-mortality group versus non-30-day-mortality group.

ELIGIBILITY:
Inclusion criteria:

1. elderly (older than 80 years old)
2. acute ischemic stroke in anterior circulation
3. NIHSS more than 8

Exclusion Criteria:

1. posterior infarction
2. ASPECT score less than 3

Ages: 80 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 1. elderly (older than 80 years old)
  2. acute ischemic stroke in anterior circulation
  3. NIHSS more than 8
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
30 days mortality | 30 days
  Patient who died in the 30 days after receiving mechanical thrombectomy

SECONDARY OUTCOMES:
The cause of mortality | 30 days
  Analyse the main cause of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Hsiang Peng, MD, Principal Investigator — FEMH
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan